CLINICAL TRIAL: NCT04529226
Title: A Randomized, Multicenter Clinical Trial to Assess the Efficacy and Safety of Clozapine vs Treatment as Usual for Treatment-resistant Psychosis in Adolescents and Young Adults With Intellectual Disability.
Brief Title: Study to Compare Clozapine vs Treatment as Usual in People With Intellectual Disability & Treatment-resistant Psychosis
Acronym: CLOZ-AID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOZ-AID; 2020-000091-37 (EudraCT Number)
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Psychosis; Intellectual Disability
MeSH Terms: conditions — Psychotic Disorders; Intellectual Disability | interventions — Clozapine; Pyrantel; Haloperidol; Pimozide; Olanzapine; Risperidone; Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clozapine (Experimental): Pharmaceutical Form: Tablet Anatomical Therapeutic Chemical classification system (ATC Code): N: nervous system, N05: psycholeptic, N05A: antipsychotic, N05AH02: clozapine (N05AH02)
  Interventions: Drug: Clozapine
- Control (Active Comparator): Usual antipsychotic medication used in the treatment of treatment-resistant psychosis.
  Interventions: Drug: haloperidol, pimozide, olanzapine, risperidone, amisulpride

INTERVENTIONS:
Drug: Clozapine — Start treatment with 12.5 mg every 12 hours with the recommendation to increase dosage by 25-50 mg/day provided it is well tolerated up to a level of 300-450 mg/day at the end of the second week
  Other Names: Nemex; Leponex
  Arms: Clozapine
Drug: haloperidol, pimozide, olanzapine, risperidone, amisulpride — Treatment as usual using first-generation or second-generation antipsychotics
  Arms: Control

SUMMARY:
This clinical trial will prove whether a large number of people with intellectual disability and treatment-resistant psychosis could benefit from the use of clozapine. Benefit will mean a measurable significant improvement in subjects' clinical response and quality of life.

DETAILED DESCRIPTION:
Randomized, open-label, multicenter phase II clinical trial that seeks to evaluate the safety and efficacy of clozapine versus standard clinical treatment in patients between the ages of 16 and 55 with intellectual disability and treatment-resistant psychosis.

Clozapine is the most effective antipsychotic for patients with non-affective psychosis who do not respond to other first and second generation antipsychotic treatments. In addition, it has been shown to be very effective in another series of clinical situations such as hostility and aggressiveness, polydipsia and in behavioral disorders and psychosis, frequent situations in people with intellectual disabilities.

The primary objective is to assess the efficacy and safety of clozapine versus standard clinical practice treatment in patients with intellectual disability and resistant psychotic disorder, as measured by change in Clinical Global Impression: Clinical Global Impression-Schizophrenia scale (ICG-SCH) global score over trial visits.

The study determines to reach a sample size of 114 patients distributed among the 25 active centers. Randomization is 1:1 and consists of 6 visits to the center spread over 12 months. At each visit, the patient will undergo a physical examination and sample collection, along with a clinical and cognitive evaluation using the scales provided in accordance with the clinical guidelines.

In addition, if the patient falls into the experimental arm (Clozapine), it is necessary to collect a blood sample weekly during the first 18 weeks and biweekly until completing the 12 months of the study, so that the medical team has special control in the analytical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 16 and 55 years
* Diagnosis of intellectual disability according to the Diagnostic and Statistical Manual of Mental Disorders Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (confirmed by a Intelligence Quotient (IQ) Score between 35 and 70 in the Kaufman test)
* Diagnosis of psychosis according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (confirmed by clinical interview).
* Treatment Resistant to antipsychotic drugs except clozapine.
* Behavioural disturbances and self-injurious behaviour over the last 6 months.
* Written informed consent of patients or legal representative.
* Negative pregnancy test (if apply)

Exclusion Criteria:

* Leukocytes < 3500/mm3 and neutrophils < 2000/mm3.
* Hypersensitivity to clozapine or excipients.
* Myeloproliferative disorders
* Uncontrolled epilepsy in the last 2 years.
* Paralytic ileus in the last 3 months.
* Diagnosis of an autism spectrum disorder
* Pregnancy and breastfeeding
* Any diseases with clozapine contraindicated.
* Any uncontrolled serious condition
* Need of treatment with more than one antipsychotic drug or electroconvulsive therapy
* Treatment with quinolones, drugs that cause agranulocytosis or drugs that affect the cytochrome P-450 enzymes.
* Risk of suicide based on the Columbia-Suicide Severity Rating Scale

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement based on Clinical Global Impression-Schizophrenia (CGI-SCH) scale score. | Baseline and 12 Months
  Overall Severity of Illness as measured by change from baseline to last study visit score
  Minimum value = 1 Normal, not ill Maximum value = 7 Among the most severely ill

SECONDARY OUTCOMES:
Clinical improvement based on Positive and Negative Syndrome Scale (PANSS) | Baseline and 12 Months
  Clinical improvement as measured by change from baseline to last study visit score
  Subjects rated from 1 to 7 on 30 different symptoms (items). Positive scale 7 Items. minimum score = 7, maximum score = 49 Negative scale 7 Items. minimum score = 7, maximum score = 49 General Psychopathology scale 16 Items. minimum score = 16, maximum score = 112
  PANSS Total score minimum = 30, maximum = 210
Clinical improvement based on Scale for the Assessment of Negative Symptoms (SANS) | Baseline and 12 Months
  Clinical improvement as measured by change from baseline to last study visit score.
  SANS is split into 5 domains, and within each domain separate symptoms are rated through a 6-point scale from 0 (absent) to 5 (severe).
  SANS Total score minimum = 0, maximum = 125
Quality of Life Improvement based on the 5 levels Quality of Life 5 dimensional (5D) 5 levels (5L) questionnaire (Euro-QoL 5D-5L scale) | Baseline and 12 Months
  Generic health status improvement measured by change from baseline to last study visit scores
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 28 days after the last investigational medicinal product administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo Facorro, Professor, Principal Investigator — Andalusian Health Service
Locations (20):
- Spain (20):
  - Unidad de Salud Mental Comunitaria Andújar, Andújar
  - Centro psicopedagógico Reina Sofía, Armilla
  - Unidad de Salud Mental Comunitaria Cabra, Cabra
  - Residencia Rodríguez Penalva, Castril
  - Hospital Universitario Reina Sofía, Córdoba
  - Unidad de Salud Mental Comunitaria Córdoba Sur, Córdoba
  - Fundación Purísima Concepción Hermanas Hospitalarias, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Residencia de Adultos María Dacia González Gordón, Jerez de la Frontera
  - Residencia para personas con Discapacidad intelectual Gravemente Afectadas Vista Hermosa, Jerez de la Frontera
  - Centro Asistencial San Juan de Dios, Málaga
  - Hospital Regional Universitario, Málaga
  - Unidad de Salud Mental Comunitaria Montilla, Montilla
  - Unidad de Salud Mental Comunitaria Montoro, Montoro
  - Villablanca Serveis Assistencials, Reus
  - Residencia de gravemente afectados Virgen de la Caridad, Sanlúcar de Barrameda
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Centro Ocupacional El Curtido, Ubrique

REFERENCES:
- [Derived] Alemany-Navarro M, Sanchez-Barbero B, Reguera-Pozuelo P, Altea-Manzano L, Gomez-Garrido A, Rocha-Gonzalez I, Garrido-Torres N, Ruiz-Veguilla M, Garcia-Cerro S, Rosso-Fernandez CM, Villagran-Moreno JM, Sarramea F, Cervilla-Ballesteros J, Martinez-Leal R, Mayoral-Cleries F; CLOZ-AID Group; Crespo-Facorro B. Efficacy of clozapine versus standard treatment in adult individuals with intellectual disability and treatment-resistant psychosis (CLOZAID): study protocol of a multicenter randomized clinical trial. Front Psychiatry. 2024 May 14;15:1400621. doi: 10.3389/fpsyt.2024.1400621. eCollection 2024. PMID 38807685